CLINICAL TRIAL: NCT04495101
Title: A Multicenter, Randomized, Open-label, Parallel Group Pilot Study to Evaluate the Safety and Efficacy of Prolastin Plus Standard Medical Treatment (SMT) Versus SMT Alone in Hospitalized Subjects With COVID-19
Brief Title: Study to Evaluate the Safety and Efficacy of Prolastin in Hospitalized Subjects With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC2005; 2020-001953-36 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: Coronavirus disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolastin 120 mg/kg + Standard Medical Treatment (Experimental): Subjects will receive Prolastin, two intravenous infusion (IV) doses of 120 milligram per kilogram (mg/kg), based upon the subject's body weight, on Day 1 and Day 8. Subjects will also receive all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Biological: Prolastin; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Subjects will receive all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: Prolastin — Intravenous infusion 120 mg/kg
  Other Names: Alpha1-proteinase inhibitor
  Arms: Prolastin 120 mg/kg + Standard Medical Treatment
Drug: Standard Medical Treatment — Standard medical treatment per local policies or guidelines
  Other Names: SMT

SUMMARY:
The primary objective of the study is to determine if Prolastin plus SMT can reduce the proportion of subjects dying or requiring intensive care unit (ICU) admission on or before Day 15 or who are dependent on invasive mechanical ventilation on Day 15 versus SMT alone in hospitalized subjects with Coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized male or female subject ≥ 18 years of age at the time of Screening who is being treated for COVID-19. Subjects must be screened within 48 hours (≤ 48 hours) of hospital admission.
2. Has laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by qualitative Polymerase Chain Reaction (PCR) (reverse transcriptase [RT]-PCR) or other commercial or public health assay in any specimen during the current hospital admission prior to randomization.
3. COVID-19 illness (symptoms) of any duration, including both of the following:

   1. Radiographic infiltrates by imaging (chest X-Ray, computerized tomography (CT) scan, etc.) and/or clinical assessment (evidence of rales/crackles on the exam) with peripheral oxygen saturation by pulse oximetry (SpO2) <94% on room air
   2. Any One of the following related to COVID-19: i. Ferritin > 400 nanogram per milliliter (ng/mL), ii. Lactate dehydrogenase (LDH) > 300 units per liter (U/L), iii. D-Dimers > reference range, or iv. C-reactive protein (CRP) > 40 milligram per liter (mg/L)
4. Subjects provides informed consent prior to the initiation of any study procedures.

Exclusion Criteria:

1. Subjects requiring invasive mechanical ventilation or ICU admission or with PaO2/FIO2 ≤ 150 mm Hg (ie, arterial oxygen in mm Hg divided by fraction inspired oxygen concentration [eg, 0.21 for room air]).
2. Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may place the subject at undue medical risk.
3. The subjects have had a known serious anaphylactic reaction to blood, any blood-derived or plasma product, or known selective immunoglobulin A (IgA) deficiency with anti-IgA antibodies.
4. A medical condition in which the infusion of additional fluid is contraindicated.
5. Shock that is unresponsive to fluid challenge and/or multiple vasopressors and accompanied by multiorgan failure considered not able to be reversed by the Principal Investigator.
6. Known alpha-1 antitrypsin deficiency for which the subject is already receiving alpha1-proteinase inhibitor augmentation therapy.
7. Women who are pregnant or breastfeeding. Female subjects of child-bearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at Screening/Baseline Visit.
8. Subjects for whom there is limitation of therapeutic effort such as "Do not resuscitate" status.
9. Currently participating in another interventional clinical trial with investigational medical product or device.
10. Subjects previously requiring long-term oxygen therapy (home oxygen therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects Dying or Requiring ICU Admission | Up to Day 15
Percentage of Subjects Who are Dependent on Invasive Mechanical Ventilation | Day 15

SECONDARY OUTCOMES:
Change from Baseline in National Early Warning Score (NEWS) | Day 1 through Day 29
Time to Clinical Response as Assessed by: NEWS ≤ 2 Maintained for 24 hours | Day 1 through Day 29
Time to Hospital Discharge | Day 1 through Day 29
Duration of ICU Stay | Up to Day 29
Duration of Any Oxygen Use | Day 1 through Day 29
Duration of Mechanical Ventilation | Up to Day 29
Mean Change from Baseline in Ordinal Scale | Day 1 through Day 29
Absolute Value Change from Baseline in Ordinal Scale | Day 1 through Day 29
Percentage of Subjects in Each Severity Category of the 7-Point Ordinal Scale | Day 15, Day 29
Time to Sustained Normalization of Temperature | Day 1 through Day 29
Percentage of Subjects who Sustained Normalization of Temperature | Day 1 through Day 29
Number of Subjects who Develop Acute Respiratory Distress Syndrome (ARDS) | Up to Day 29
Length of Time to Clinical Progression | Up to Day 29
Mortality Through Day 29 | Up to Day 29

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No